CLINICAL TRIAL: NCT04765774
Title: The Effect of Expressive Touch and Music Applied After Lumbar Disc Hernia Surgery on Pain, Vital Signs, and Near-infrared Spectroscopy (NIRS) Values.
Brief Title: The Effect of Expressive Touch and Music Applied After Lumbar Disc Hernia Surgery.
Acronym: NIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Neslihan SÖYLEMEZ, research assistant, Inonu University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: InonuUniversity
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Lumbar Disc Herniation
Keywords: Nursing; Touch; Music; Pain; Near-İnfrared Spectroscopy
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Effect of Expressive Touch Applied After Lumbar Disc Herniation Surgery (Experimental): Expressive touch reduces pain and keeps vital signs and NIRS values within normal limits by touching the arms and hands of the patients through energy transfer.
  Interventions: Other: Ekspressive touch
- The Effect of Music Applied After Lumbar Disc Herniation Surgery (Experimental): Patients listening to music are distracted and their pain is reduced, vital signs and NIRS values are kept within normal limits.
  Interventions: Other: Music
- Pain, vital signs and NIRS values of patients after lumbar disc hernia surgery (No Intervention): No intervention is applied to the patients in this group and the effectiveness of the interventions used on the patients in the other group is measured.

INTERVENTIONS:
Other: Ekspressive touch — Patients will be divided into three groups. The expressive touch group will touch the patient's hand.
  Arms: The Effect of Expressive Touch Applied After Lumbar Disc Herniation Surgery
Other: Music — The music chosen by the patient will be played in the music group.
  Arms: The Effect of Music Applied After Lumbar Disc Herniation Surgery

SUMMARY:
Patients undergoing lumbar hernia surgery will be divided into expressive touch, music and control groups. Pre-test and post-test pain levels, vital signs, and NIRS values of the patients will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* General anesthesia applied,
* Patients with the same type of treatment protocol,
* Verbal pain score with at least 4,
* Patients with a Ramsay sedation Scale score of 3 and below,
* Without a chronic disease,
* Without a disease (AVM, blockage of brain vessels, etc.) that will affect brain oxygenation,
* Who has not been diagnosed with any psychiatric illness
* No hearing and perception problems,
* No loss of sensation in upper extremity according to light touch test,
* Any complications after surgery are undeveloped

Exclusion Criteria:

* Do not meet the inclusion criteria,
* Interrupting the research,
* Patients with incomplete answers to questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Expressive touch applied to patients with lumbar disc herniation surgery reduces the level of pain. | 30 minute
  the patient relaxes as a result of expressive touch, pain value will be measured by the verbal pain scale. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery doesn't reduce the level of pain. | 30 minute
  the patient doesn't relaxes as a result of expressive touch, pain value will be measured by the verbal pain scale. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Music applied to patients with lumbar disc hernia surgery reduces the level of pain. | 30 minute
  the patient relaxes as a result of music. the verbal pain scale will be measured pain value. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Music applied to patients with lumbar disc hernia surgery doesn't reduce the level of pain. | 30 minute
  the patient doesn't relax as a result of music. the verbal pain scale will be measured pain value. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery is more effective than music in reducing pain. | 30 minute
  the patient doesn't relax as a result of music but relaxes by expressive touch. The verbal pain scale will be measured pain value. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery is not more effective than music in reducing pain. | 30 minute
  the patient doesn't relax as a result of expressive touch but relaxes by music. The verbal pain scale will be measured pain value. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery ensures that body temperature, pulse, respiratory rate, blood pressure, and saturation values are kept within physiological limits. | 1 and a half hours
  the patient relaxes as a result of expressive touch. Body temperature will be measured with a digital thermometer. Pulse and blood pressure value will be measured with a digital sphygmomanometer. The respiratory rate will be calculated by counting. Oxygen saturation will be measured by pulse oximetry. The initiative will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery doesn't affect body temperature, pulse, respiratory rate, blood pressure and saturation values within physiological limits. | 1 and a half hours
  the patient doesn't relax as a result of expressive touch. Body temperature will be measured with a digital thermometer. Pulse and blood pressure value will be measured with a digital sphygmomanometer. The respiratory rate will be calculated by counting. Oxygen saturation will be measured by pulse oximetry. The initiative will be evaluated 3 times. 44 patients will be measured in the touch group.
Music applied to patients with lumbar disc herniation surgery ensures that body temperature, pulse, respiratory rate, blood pressure, and saturation values are kept within physiological limits. | 1 and a half hours
  the patient relaxes as a result of music. Body temperature will be measured with a digital thermometer. Pulse and blood pressure value will be measured with a digital sphygmomanometer. The respiratory rate will be calculated by counting. Oxygen saturation will be measured by pulse oximetry. The initiative will be evaluated 3 times. 44 patients will be measured in the touch group.
Music applied to patients with lumbar disc herniation surgery doesn't affect body temperature, pulse, respiratory rate, blood pressure, and saturation values are kept within physiological limits. | 1 and a half hours
  the patient doesn't relax as a result of music. Body temperature will be measured with a digital thermometer. Pulse and blood pressure value will be measured with a digital sphygmomanometer. The respiratory rate will be calculated by counting. Oxygen saturation will be measured by pulse oximetry. The initiative will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery is more effective than music in keeping body temperature, pulse, respiratory rate, blood pressure, and saturation values are within physiological limits. | 1 and a half hours
  the patient doesn't relax as a result of music but relaxes by expressive touch. Body temperature will be measured with a digital thermometer. Pulse and blood pressure value will be measured with a digital sphygmomanometer. The respiratory rate will be calculated by counting. Oxygen saturation will be measured by pulse oximetry. The initiative will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery is not more effective than music in keeping body temperature, pulse, respiratory rate, blood pressure, and saturation values are within physiological limits. | 1 and a half hours
  the patient doesn't relax as a result of expressive touch but relaxes by music. Body temperature will be measured with a digital thermometer. Pulse and blood pressure value will be measured with a digital sphygmomanometer. The respiratory rate will be calculated by counting. Oxygen saturation will be measured by pulse oximetry. The initiative will be evaluated 3 times. 44 patients will be measured in the touch group.
The expressive touch applied to patients with lumbar disc herniation surgery increases the Near Infrared Spectroscopy (NIRS) value. | 30 minute
  the patient relaxes as a result of expressive touch. NIRS value will be measured by a digital measuring device. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
The expressive touch applied to patients with lumbar disc herniation surgery doesn't increase the Near Infrared Spectroscopy (NIRS) value. | 30 minute
  the patient doesn't relax as a result of expressive touch. NIRS value will be measured by a digital measuring device. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
The music applied to patients with lumbar disc herniation surgery increases the Near Infrared Spectroscopy (NIRS) value. | 30 minute
  the patient relaxes as a result of music. NIRS value will be measured by a digital measuring device. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
The music applied to patients with lumbar disc herniation surgery doesn't increase the Near Infrared Spectroscopy (NIRS) value. | 30 minute
  the patient doesn't relax as a result of music. NIRS value will be measured by a digital measuring device. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery is more effective than music in increasing NIRS values. | 30 minute
  the patient doesn't relax as a result of music but relaxes by expressive touch. NIRS value will be measured by a digital measuring device. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.
Expressive touch applied to patients with lumbar disc herniation surgery is not more effective than music in increasing NIRS values. | 30 minute
  the patient doesn't relax as a result of expressive touch but relaxes by music. NIRS value will be measured by a digital measuring device. The attempt will be evaluated 3 times. 44 patients will be measured in the touch group.

CONTACTS AND LOCATIONS:
Overall Officials: meral özkan, PhD, Principal Investigator — Inonu University
Locations (1):
- İnonu University, Battalgazi, Malatya, Turkey (Türkiye)